CLINICAL TRIAL: NCT03045120
Title: Determining Change in Cardiovascular and Metabolic Risks in Patients With Chronic Phase Chronic Myeloid Leukemia Receiving BCR-ABL Tyrosine Kinase Inhibitor First-Line Therapy in the United States
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA180-653
Record Dates: First submitted 2017-01-31; First posted 2017-02-07 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Chronic Phase Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biomarker analyses will be collected for metabolic panels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- dasatinib cohort: Intended to characterize the impact of dasatinib on cardiovascular and metabolic risk factors in CP-CML treated patients who are TKI naive and initiating first line TKIs in routine clinical practice in the US.
- imatinib cohort: Intended to characterize the impact of imatinib on cardiovascular and metabolic risk factors in CP-CML treated patients who are TKI naive and initiating first line TKIs in routine clinical practice in the US.
- nilotinib cohort: Intended to characterize the impact of nilotinib on cardiovascular and metabolic risk factors in CP-CML treated patients who are TKI naive and initiating first line TKIs in routine clinical practice in the US.
- bosutinib cohort: Intended to characterize the impact of bosutinib on cardiovascular and metabolic risk factors in CP-CML treated patients who are TKI naive and initiating first line TKIs in routine clinical practice in the US.

SUMMARY:
This non-interventional, prospective study will characterize the impact of three approved first and second generation BCR-ABL1 tyrosine kinase inhibitors on cardiovascular and metabolic risk factors in chronic phase CML (CP-CML) patients who are TKI naive and initiating first-line TKIs in routine clinical practice in the US. All treatment decisions will be determined at the discretion of the treating physician(s) and data identifying the cardiovascular and metabolic risk factors will be collected. Additional fasting blood samples (collected following 8 hours of fasting) will be collected during standard of care (SOC)/routine office visits. Additional research imaging will be performed and will be reviewed by core imaging laboratory. As the study is collecting data on management of CML, this study will not influence the prescribing or management practices at participating sites.

DETAILED DESCRIPTION:
This non-interventional, prospective study will characterize the impact of three approved first and second generation BCR-ABL1 tyrosine kinase inhibitors on cardiovascular and metabolic risk factors in chronic phase CML (CP-CML) patients who are TKI naive and initiating first-line TKIs in routine clinical practice in the US. All treatment decisions will be determined at the discretion of the treating physician(s) and data identifying the cardiovascular and metabolic risk factors will be collected. Additional fasting blood samples (collected following 8 hours of fasting) will be collected during standard of care (SOC)/routine office visits. Additional research imaging will be performed and will be reviewed by core imaging laboratory. As the study is collecting data on management of CML, this study will not influence the prescribing or management practices at participating sites.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years at the time of Ph+ CP-CML diagnosis
2. Newly diagnosed chronic phase of Ph+ CP-CML, confirmed with cytogenetic and/or molecular testing at baseline
3. Treatment-naïve and initiating treatment with dasatinib, imatinib, nilotinib or bosutinib
4. Willingness and ability to comply with routine office visits

Exclusion Criteria:

1. Any other prior or active non-CML active malignancy for which the patient is receiving treatment
2. Participation in a therapeutic clinical trial for CML disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly-diagnosed, treatment-naïve CP-CML patients who are ≥ 18 years at the time of CP-CML diagnosis who are scheduled to initiate treatment with dasatinib, imatinib, nilotinib or Bosutinib are eligible for enrollment. Enrolled patients (n=200) will be distributed across the 3 patient treatment groups of newly diagnosed CP-CML patients who will initiate their first- line TKI treatment
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
changes in cardiovascular risk from baseline using the Framingham Coronary Heart Disease Score | up to 24 months
changes in metabolic risk from baseline using metabolic lab values | up to 24 months

SECONDARY OUTCOMES:
echocardiography to assess left ventricular function | up to 24 months
urinary protein excretion to assess early vascular endothelial changes | up to 24 months
coronary calcium scoring to assess coronary artery narrowing | up to 24 months
metabolic labs (Plasma Glucose, HbA1c, Fasting Lipids) for assessing the metabolic disease | up to 24 months
safety and tolerability of first-line BCR-ABL TKIs in adults with CP-CML based on the number of treatment-related adverse events collected in the medical records | up to 24 months
clinical outcomes as described by the number of deaths from clinical assessments of disease status and mutational analysis | up to 24 months
clinical outcomes as described by the major molecular response from clinical assessments of disease status and mutational analysis | up to 24 months
clinical outcomes as described by the cytogenetic response from clinical assessments of disease status and mutational analysis | up to 24 months
time to development of clinical outcomes from baseline to time of clinical outcome event based on clinical assessments | up to 24 months
description of treatment patterns based on the number of changes in treatment dosing, interruptions, changes in therapy, duration of therapy and treatment discontinuations through the management of adverse events and comorbid disease | up to 24 months
description of the demographic and clinical patient characteristics associated with initial treatment choice and changes of treatment based on the medical records | up to 24 months
measurement of serum biomarkers that are predictive of an increased risk for cardiovascular or metabolic disease | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- United States (24):
  - Mount Sinai Hospital, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - The Cancer Institute At Alexian Brothers, Elk Grove Village, Illinois
  - Northwest Oncology & Hematology, SC, Hoffman Estates, Illinois
  - Hematology/Oncology Of The North Shore, Lake Forest, Illinois
  - Northwest Oncology & Hematology, SC, Rolling Meadows, Illinois
  - Healthcare Research Network III, LLC, Tinley Park, Illinois
  - American Health Network, Avon, Indiana
  - Cancer Center Of Kansas, Wichita, Kansas
  - Hazard Arh Regional Medical Center, Hazard, Kentucky
  - St. Agnes Hospital, Baltimore, Maryland
  - St Vincent Frontier Cancer Center, Billings, Montana
  - Local Institution - 0009, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Med Col Of Cornell, New York, New York
  - Columbia University Medical Center (Cumc), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Leo W.Jenkins Cancer Center, Greenville, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - Providence Regional Cancer Partnership, Everett, Washington
  - Fred Hutchinson Can Res Ctr, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Educational Resource — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: EAP Investigator Requests — http://www.bms.com/clinical_trials/investigator_sponsored_research/Pages/expanded-access-program.aspx